CLINICAL TRIAL: NCT03865251
Title: Effects of Kinesiology Tape Tensions on Gastrocnemius and Soleus H-reflex Modulations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Taipei (Other)
Responsible Party: Principal Investigator, YUNG-SHENG CHEN, Associate Professor, University of Taipei
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: UTaipei
Record Dates: First submitted 2019-03-01; First posted 2019-03-06 (Actual); Last update posted 2020-07-30 (Actual); Status verified 2020-07

CONDITIONS: Kinesiology Taping
Keywords: H-reflex modulation; motoneuronal excitability; Ia afferent inputs; posture; Kinesiology tape

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- experimental group (Experimental): Kinesiology tape application to dominant leg during lying and standing positions
  Interventions: Device: Kinesiology tape

INTERVENTIONS:
Device: Kinesiology tape — Application for 0%, 50%, and 100% of maximal KT stretch to the calf muscle during lying and standing positions

SUMMARY:
Kinesio tape (KT) has been widely used in the areas of sports and physical therapy (Kase, 2003). The effect of KT tensions on H-reflex modulation has not been discussed in the literature. This study investigated the effect of different KT tensions on the H-reflex modulation in the gastrocnemius and the soleus muscles.

ELIGIBILITY:
Inclusion Criteria:

* Undertake regular exercise at least 3 times a week with accumulation of 150 min per week
* Age between 20 and 30 years old

Exclusion Criteria:

* History of severe neuromuscular injury
* Current lower extremity injury
* Current neurological diseases

Ages: 20 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2019-02-18 (Actual); Primary Completion 2019-04-15 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
H-reflex and M-wave ratio | 30 min before kinesiology taping application
  Electromyographic record
H-reflex and M-wave ratio | During kinesiology taping application
  Electromyographic record
H-reflex and M-wave ratio | Immediately following kinesiology taping application
  Electromyographic record

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Exercise and Health Sciences, University of Taipei, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided